CLINICAL TRIAL: NCT02349698
Title: A Clinical Research of Chimeric Antigen Receptor (CAR) T Cells Targeting CD19 Positive Malignant B-cell Derived Leukemia and Lymphoma
Brief Title: A Clinical Research of CAR T Cells Targeting CD19 Positive Malignant B-cell Derived Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shiqi Li, Researcher of Biotherpy Center, Southwest Hospital, China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-001
Record Dates: First submitted 2015-01-25; First posted 2015-01-29 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Leukemia; Lymphoma
Keywords: CAR T; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acute Lymphoblastic Leukemia (Other): Acute lymphoblastic leukemia treated with chimeric antigen receptor modified T cells targeting CD19.
  Interventions: Biological: Chimeric Antigen Receptor Modified T cells Targeting CD19
- Chronic Lymphcytic Leukemia (Other): Chronic lymphocytic leukemia with chimeric antigen receptor modified T cells targeting CD19.
  Interventions: Biological: Chimeric Antigen Receptor Modified T cells Targeting CD19
- Non-Hodgkin Lymphoma (Other): Non-hodgkin lymphoma treated with chimeric antigen receptor modified T cells targeting CD19.
  Interventions: Biological: Chimeric Antigen Receptor Modified T cells Targeting CD19

INTERVENTIONS:
Biological: Chimeric Antigen Receptor Modified T cells Targeting CD19 — T cells modified with CD19 targeted chimeric antigen receptor.

SUMMARY:
The main purpose of this research is to verify the safety of CD19 targeted chimeric antigen receptor T cells and to determine the proper dosage of CAR T cells infused.

DETAILED DESCRIPTION:
Nowadays refractory or relapsed leukemia/lymphoma lacks effective treatment. Innovative therapy is urgently required. Chimeric antigen receptor (CAR)-modified T cells have demonstrated great successes in treating even late stage cluster of differentiation antigen 19 (CD19) positive B cell malignancies. To design better CAR T cells, we have developed new CD19 CARs. Preclinical studies have demonstrated effective killing of CD19 target cells. In this study, the CD19 CARs, will be evaluated in CD19 positive leukemia/lymphoma patients. The primary goal is to confirm its adverse effects including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell derived acute lymphoblastic leukemia(ALL), chronic lymphocytic leukemia(CLL) and non-hodgkin lymphoma.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 4 years to 75 years.
5. Disease progresses but reserves reaction to recent treatments.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.

Exclusion Criteria:

1. HIV affected.
2. Patients are allergic to cytokines.
3. Central nervous system leukemia within 28 days.
4. Uncontrolled active infection.
5. Acute or chronic GVHD.
6. Treated with T cell inhibitor.
7. Pregnancy and nursing females.
8. Other situations we think improper for the research.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events of each patient. | 3 years
  Determine the toxicity profile of the CD19 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-CD19 CAR T cells in vivo. | 3 years
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Efficacy of anti-CD19 CAR T cells assessed by the ability of CAR T cells to kill leukemia/lymphoma cells | 12 weeks
Maximum tolerated dose (MTD) of CD19 targeted CAR T cells. | 4 weeks
  To confirm the maximum tolerated dose of CD19 targeted CAR T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD, PhD, Study Chair — Biotherapy Center of Southwest Hospital
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Htun KT, Gong Q, Ma L, Wang P, Tan Y, Wu G, Chen J. Successful Treatment of Refractory and Relapsed CNS Acute Lymphoblastic Leukemia With CD-19 CAR-T Immunotherapy: A Case Report. Front Oncol. 2021 Aug 26;11:699946. doi: 10.3389/fonc.2021.699946. eCollection 2021. PMID 34513679
- [Derived] Heng G, Jia J, Li S, Fu G, Wang M, Qin D, Li Y, Pei L, Tian X, Zhang J, Wu Y, Xiang S, Wan J, Zhu W, Zhang P, Zhang Q, Peng X, Wang L, Wang P, Wei Z, Zhang Y, Wang G, Chen X, Zhang C, Sun Y, Zhao W, Fan Y, Yang Z, Chen J, Qian C. Sustained Therapeutic Efficacy of Humanized Anti-CD19 Chimeric Antigen Receptor T Cells in Relapsed/Refractory Acute Lymphoblastic Leukemia. Clin Cancer Res. 2020 Apr 1;26(7):1606-1615. doi: 10.1158/1078-0432.CCR-19-1339. Epub 2019 Nov 15. PMID 31732519